CLINICAL TRIAL: NCT01784211
Title: The Pharmacokinetic and Pharmacodynamic Intra-subject Variability of LY2605541 and the Effect of Exercise on LY2605541 Pharmacokinetics in Patients With Type 1 Diabetes Mellitus
Brief Title: A Study of LY2605541 and Glargine and Exercise in Participants With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14183; I2R-MC-BIAW (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-02-01; First posted 2013-02-05 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — LY2605541; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- LY2605541 (Part A) (Experimental): 0.5 units per kilogram (U/kg) LY2605541 subcutaneously (SC) once daily for 15 days. Part A involved 3 clamp procedures on Days 8, 11, and 14. Participants remained on their regular physician-prescribed mealtime insulin.
  Interventions: Drug: LY2605541
- Glargine (Part A) (Active Comparator): 0.5 U/kg insulin glargine SC once daily for 15 days. Part A involved 3 clamp procedures on Days 8, 11, and 14. Participants remained on their regular physician-prescribed mealtime insulin.
  Interventions: Drug: Insulin Glargine
- First LY2605541 + Exercise,Then LY2605541 Alone (Part B) (Experimental): 0.5 U/kg LY2605541 SC once daily for an additional 6 days, beginning on Day 16. Exercise challenge on Day 17 (no exercise on Day 20).Participants remained on their regular physician-prescribed mealtime insulin.
  Interventions: Drug: LY2605541
- First LY2605541 Alone, Then LY2605541 + Exercise (Part B) (Experimental): 0.5 U/kg LY2605541 SC once daily for an additional 6 days, beginning on Day 16. Exercise challenge on Day 20 (no exercise on Day 17). Participants remained on their regular physician-prescribed mealtime insulin.
  Interventions: Drug: LY2605541
- First Glargine + Exercise, Then Glargine Alone (Part B) (Active Comparator): 0.5 U/kg insulin glargine SC once daily for an additional 6 days, beginning on Day 16. Exercise challenge on Day 17 (no exercise on Day 20). Participants remained on their regular physician-prescribed mealtime insulin.
  Interventions: Drug: Insulin Glargine
- First Glargine Alone, Then Glargine + Exercise (Part B) (Active Comparator): 0.5 U/kg insulin glargine SC once daily for an additional 6 days, beginning on Day 16. Exercise challenge on Day 20 (no exercise on Day 17).
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: LY2605541
  Arms: First LY2605541 + Exercise,Then LY2605541 Alone (Part B); First LY2605541 Alone, Then LY2605541 + Exercise (Part B); LY2605541 (Part A)
Drug: Insulin Glargine
  Arms: First Glargine + Exercise, Then Glargine Alone (Part B); First Glargine Alone, Then Glargine + Exercise (Part B); Glargine (Part A)

SUMMARY:
The purpose of this study is to measure how much of the study drug or insulin glargine gets into the blood stream and how long it takes the body to get rid of it. The effect of exercise will also be evaluated.

This study has two parts. In Part A, each participant will receive a daily injection of LY2605541 or insulin glargine for about 15 days. Some participants may continue into Part B. In Part B, participants will receive a daily injection of LY2605541 or insulin glargine with or without exercise. Part B lasts about 6 days.

Participants will remain on their regular physician-prescribed mealtime insulin throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Are males or females that have had a diagnosis of Type I Diabetes Mellitus (T1DM) for at least 12 months and are receiving multiple daily insulin injections. Total daily insulin dose <1.2 units per kilogram per day (U/kg/day); daily basal dose >0.2 U/kg/day
* Female participants: are women of child-bearing potential who test negative for pregnancy at the time of enrollment based on a urine pregnancy test and agree to use a reliable method of birth control during the study
* Have a body mass index (BMI) of 18 to 30 kilograms per meter squared (kg/m^2), inclusive
* Have a fasting c-peptide <0.3 nanomoles per liter (nmol/L)
* Have a hemoglobin A1c (HbA1c) <9% at screening

Participants with T1DM are eligible for enrollment in Part B of the study only if they meet all of the following criteria:

* Have a maximal oxygen uptake (VO2 max) of ≥25 milliliters (mL) of oxygen per kilogram per minute (O2/kg/min) (for women) or ≥30 mL O2/kg/min (for men)
* Perform regular physical cardiorespiratory activity to achieve an average total energy expenditure of ≥500 metabolic equivalent of task (MET)-minutes per week during the last 3 months prior to screening

Exclusion Criteria:

* Have known allergies to LY2605541, insulin glargine, related compounds or any components of the formulation
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine (apart from T1DM), hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Have had episodes of severe hypoglycemia in the past 6 months (severe hypoglycemia is defined as having neurological symptoms consistent with neuroglycopenia and having required assistance in treatment by a second party)
* Have a history of hypoglycemia unawareness
* Regular use or intended use of any over-the-counter or prescription medications or nutritional supplements that may affect blood glucose, the body's sensitivity to insulin, or that promote weight loss within 14 days prior to dosing
* Have an average weekly alcohol intake that exceeds 21 units per week (males up to age 65) and 14 units per week (males over 65 and females), or are unwilling to comply with study requirements regarding alcohol consumption
* Currently smokes >5 cigarettes per day, or are unwilling to comply with study requirements regarding smoking or use of tobacco products
* Have a hemoglobin level <8.0 millimoles per liter (mmol/L) (male) or <6.4 mmol/L (female) at screening
* Are currently participating in a weight loss program or plan to do so during the course of the study
* Are receiving chronic (lasting longer than 14 consecutive days) systemic glucocorticoid therapy (excluding topical, intra-articular, and intra-ocular preparations) or have received such therapy within the 4 weeks before dosing
* Have fasting triglycerides >400 milligrams per deciliter (mg/dL) (4.52 mmol/L)
* Have previous history or family history of deep vein thrombosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neuss, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part A is 2- arm parallel open label.
  Part B is a crossover study with 2 treatment arms (LY2605541 & Glargine), each treatment arm consists of 2 sequences.
  Sequence 1: participants received treatment on days 16,17,18,19 & 20 with exercise on day 17.
  Sequence 2: participants received treatment on days 16,17,18,19, & 20 with exercise on day 20.
Groups:
- LY2605541 (Part A): 0.5 units per kilogram (U/kg) LY2605541 subcutaneously (SC) once daily for 15 days. Part A involved 3 clamp procedures on Days 8, 11, and 14.
- Glargine (Part A): 0.5 U/kg insulin glargine SC once daily for 15 days. Part A involved 3 clamp procedures on Days 8, 11, and 14.
- First LY2605541 + Exercise, Then LY2605541 Alone (Part B): 0.5 U/kg LY2605541 SC once daily for an additional 6 days, beginning on Day 16. Exercise challenge on Day 17 (no exercise on Day 20).
- First LY2605541 Alone, Then LY2605541 + Exercise (Part B): 0.5 U/kg LY2605541 SC once daily for an additional 6 days, beginning on Day 16. Exercise challenge on Day 20 (no exercise on Day 17).
- First Glargine + Exercise, Then Glargine Alone (Part B): 0.5 U/kg insulin glargine SC once daily for an additional 6 days, beginning on Day 16. Exercise challenge on Day 17 (no exercise on Day 20).
Period: Part A (Days 1-15)
Arm/Group | LY2605541 (Part A) | Glargine (Part A) | First LY2605541 + Exercise, Then LY2605541 Alone (Part B) | First LY2605541 Alone, Then LY2605541 + Exercise (Part B) | First Glargine + Exercise, Then Glargine Alone (Part B) | First Glargine Alone, Then Glargine + Exercise (Part B)
Started | 38 | 38 | 0 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 37 | 38 | 0 | 0 | 0 | 0
Entered Part B | 19 (Participants who completed Part A and met certain criteria had the option of continuing to Part B.) | 21 (Participants who completed Part A and met certain criteria had the option of continuing to Part B.) | 0 | 0 | 0 | 0
Completed | 35 | 36 | 0 | 0 | 0 | 0
Not Completed | 3 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0 | 0 | 0
Period: Part B (Days 16-21)
Arm/Group | LY2605541 (Part A) | Glargine (Part A) | First LY2605541 + Exercise, Then LY2605541 Alone (Part B) | First LY2605541 Alone, Then LY2605541 + Exercise (Part B) | First Glargine + Exercise, Then Glargine Alone (Part B) | First Glargine Alone, Then Glargine + Exercise (Part B)
Started | 0 (Participants who completed Part A and met certain criteria had the option of continuing to Part B.) | 0 (Participants who completed Part A and met certain criteria had the option of continuing to Part B.) | 10 | 9 | 11 | 10
Completed | 0 | 0 | 10 | 9 | 11 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were randomized and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2605541 (Part A) | Glargine (Part A) | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (10.8) | 42.0 (12.1) | 42.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 11 | 15
  Male | 33 | 27 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 36 | 38 | 74
  Multiple | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 37 | 38 | 75

OUTCOME MEASURES:

1. Primary Outcome: Part A: Pharmacokinetics: Area Under the Concentration Versus Time Curve Over the Dosing Interval (AUCτ) of LY2605541 and Insulin Glargine: Intra-Participant Variability
Description: Venous blood samples for pharmacokinetic analysis were collected during the euglycemic glucose clamps during Part A. The intra-participant percentage of coefficient of variation (%CV) is presented. %CV was calculated by dividing the standard deviation by the mean, multiplied by 100.
Time Frame: Part A: Predose and 4, 8, 12, and 24 hours postdose on Days 8, 11, and 14
Population: Participants in Part A who received at least 1 dose of study drug and had evaluable AUCτ data.
Measure: Number (90% Confidence Interval); unit: %CV
Groups:
- LY2605541 (Part A): 0.5 U/kg LY2605541 SC once daily for 15 days. Part A involved 3 clamp procedures on Days 8, 11, and 14.
Arm/Group | LY2605541 (Part A) | Glargine (Part A)
Number analyzed (Participants) | 37 | 23
%CV | 11.3 [9.89 to 13.2] | 19.2 [15.5 to 25.5]

2. Primary Outcome: Part A: Pharmacokinetics: Maximum Drug Concentration (Cmax) of LY2605541 and Insulin Glargine: Intra-Participant Variability
Description: as for outcome 1
Time Frame: Part A: Predose and 4, 8, 12, and 24 hours postdose on Days 8, 11, and 14
Population: Participants in Part A who received at least 1 dose of study drug and had evaluable Cmax data.
Measure: Number (90% Confidence Interval); unit: %CV
Arm/Group | LY2605541 (Part A) | Glargine (Part A)
Number analyzed (Participants) | 37 | 35
%CV | 12.6 [11.0 to 14.7] | 27.7 [23.8 to 33.3]

3. Secondary Outcome: Part A: Pharmacodynamics: Total Amount of Glucose Infused Over the Duration of the Clamp (Gtot): Intra-Participant Variability
Description: Glucodynamic measurements were collected during the euglycemic glucose clamps during Part A. The intra-participant percentage of coefficient of variation (%CV) is presented. %CV was calculated by dividing the standard deviation by the mean, multiplied by 100.
Time Frame: Part A: Predose up to 24 hours postdose on Days 8, 11, and 14
Population: Participants in Part A who received at least 1 dose of study drug and had evaluable Gtot data.
Measure: Number (90% Confidence Interval); unit: %CV
Arm/Group | LY2605541 (Part A) | Glargine (Part A)
Number analyzed (Participants) | 37 | 37
%CV | 41.4 [36.1 to 49.0] | 63.9 [55.2 to 76.6]

4. Secondary Outcome: Part B: Pharmacokinetics: AUCτ of LY2605541 and Insulin Glargine: Exercise Versus Non-Exercise
Description: Venous blood samples for pharmacokinetic analysis were collected in Part B. Results were stratified by whether or not the participant was undergoing an exercise challenge (+ Exercise) at the time of sample collection.
Time Frame: Part B: Predose, 11 hours postdose, every 30 minutes from 16.5 to 20 hours postdose, and 24 hours postdose on Day 16 or 19
Population: Participants in Part B who received at least 1 dose of study drug and had evaluable AUCτ data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles*hour per liter (pmol*h/L)
Groups:
- LY2605541 + Exercise (Part B): 0.5 U/kg LY2605541 SC once daily for an additional 6 days. Exercise challenge on Day 17 or 20.
- LY2605541 (Part B): 0.5 U/kg LY2605541 SC once daily for an additional 6 days.
- Glargine + Exercise (Part B): 0.5 U/kg insulin glargine SC once daily for an additional 6 days. Exercise challenge on Day 17 or 20.
- Glargine (Part B): 0.5 U/kg insulin glargine SC once daily for an additional 6 days.
Arm/Group | LY2605541 + Exercise (Part B) | LY2605541 (Part B) | Glargine + Exercise (Part B) | Glargine (Part B)
Number analyzed (Participants) | 18 | 18 | 10 | 9
picomoles*hour per liter (pmol*h/L) | 147000 (25) | 130000 (23) | 2950 (24) | 2650 (23)

5. Secondary Outcome: Part B: Pharmacokinetics: Cmax of LY2605541 and Insulin Glargine: Exercise Versus Non-Exercise
Description: as for outcome 4
Time Frame: as for outcome 4
Population: Participants in Part B who received at least 1 dose of study drug and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles per liter (pmol/L)
Groups:
- LY2605541 - No Exercise (Part B): 0.5 U/kg LY2605541 SC once daily for an additional 6 days.
- Glargine - No Exercise (Part B): 0.5 U/kg insulin glargine SC once daily for an additional 6 days.
Arm/Group | LY2605541 + Exercise (Part B) | LY2605541 - No Exercise (Part B) | Glargine + Exercise (Part B) | Glargine - No Exercise (Part B)
Number analyzed (Participants) | 19 | 19 | 14 | 14
picomoles per liter (pmol/L) | 11100 (27) | 6760 (28) | 166 (51) | 153 (35)

ADVERSE EVENTS:
Description: As per planned analysis adverse events were reported per intervention irrespective of exercise/ no exercise..
Groups:
- LY2605541 (Part A and Part B): Part A: 0.5 U/kg LY2605541 SC once daily for 15 days. Part A involved 3 clamp procedures on Days 8, 11, and 14.
  Participants who completed Part A and met certain criteria had the option of continuing to Part B.
  Part B: 0.5 U/kg LY2605541 SC once daily for an additional 6 days. Exercise challenge on Day 17 or 20.
- Glargine (Part A and Part B): Part A: 0.5 U/kg insulin glargine SC once daily for 15 days. Part A involved 3 clamp procedures on Days 8, 11, and 14.
  Participants who completed Part A and met certain criteria had the option of continuing to Part B.
  Part B: 0.5 U/kg insulin glargine SC once daily for an additional 6 days. Exercise challenge on Day 17 or 20.
Arm/Group | LY2605541 (Part A and Part B) | Glargine (Part A and Part B)
Serious Adverse Events (participants affected / at risk) | 1/37 | 0/38
Other Adverse Events (participants affected / at risk) | 10/37 | 12/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2605541 (Part A and Part B) (N=37) | Glargine (Part A and Part B) (N=38)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2605541 (Part A and Part B) (N=37) | Glargine (Part A and Part B) (N=38)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 8 (14) | 7 (19)
Presyncope (Nervous system disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days